CLINICAL TRIAL: NCT00430989
Title: Large, Randomised, Parallel-group, Controlled Trial, With Patients Randomly Allocated to Either N2O-containing (70% N2O in Oxygen [FiO2 0.3]) or N2O-free (70% Nitrogen in Oxygen [FiO2 0.3]).
Brief Title: The ENIGMA II Trial:Nitrous Oxide Anaesthesia and Cardiac Morbidity After Major Surgery: a Randomised Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6/07
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Anaesthesia; Major Surgery; Coronary artery disease; Nitrous oxide; Effects of Nitrous Oxide following Anaesthesia; Anaesthesia and coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nitrous Oxide

STUDY DESIGN:
Intervention Model Description: international, randomised, assessor-blinded trial in patients aged at least 45 years with known or suspected coronary artery disease having major non-cardiac surgery.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The treating anaesthetist will be unblinded to the allocation. All other personnel (surgeon, participant and outcome assessor are all blinded to treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 70% Nitrous Oxide (Other): General anaesthesia using 70% Nitrous Oxide with fraction of inspired oxygen at 30%
  Interventions: Other: Nitrous Oxide
- No Nitrous Oxide (Other): General anaesthesia not containing Nitrous oxide with fraction of inspired oxygen at 30%
  Interventions: Other: No Nitrous Oxide

INTERVENTIONS:
Other: Nitrous Oxide — General anaesthesia with the inclusion of Nitrous Oxide at 70%
  Arms: 70% Nitrous Oxide
Other: No Nitrous Oxide — General anaesthesia with no use of Nitrous Oxide
  Arms: No Nitrous Oxide

SUMMARY:
To investigate the safety of nitrous oxide (N2O) anaesthesia in patients with risk factors for coronary artery disease undergoing major surgery.

DETAILED DESCRIPTION:
Approximately 25% of patients undergoing major surgery have known coronary artery disease (CAD) or risk factors for CAD.

N2O interferes with vitamin B12 and folate metabolism. This impairs production of methionine (from homocysteine), used to form tetrahydrofolate and thymidine during DNA synthesis. It has been repeatedly demonstrated that N2O anaesthesia increases postoperative homocysteine levels. Chronic hyperhomocysteinaemia is associated with cardiovascular disease, and acute hyperhomocysteinaemia is known to cause endothelial dysfunction. One small trial has demonstrated an increased incidence of postoperative myocardial ischaemia in patients receiving N2O anaesthesia. Reducing postoperative myocardial infarction and death are important aims for those with CAD undergoing major surgery.

Our previous trial (ENIGMA) studied 2050 patients and identified some serious adverse effects, but most patients were not at risk of CAD and so we could not reliably assess serious cardiac complications. We propose a large simple randomized clinical trial of 7,000 patients to provide a definitive evaluation of the safety of N2O anaesthesia.

Updated statistical analysis plan can be found at www.enigma2.org.au.

ELIGIBILITY:
Inclusion Criteria

1. Adult males and females age ≥ 45 years, undergoing noncardiac surgery and general anaesthesia expected to exceed two hours.
2. At increased risk of cardiac events, defined as any of

   1. history of coronary artery disease as defined by a history of any one of the following: i. angina ii. MI iii. segmental wall motion abnormality on echocardiography or a fixed defect on radionuclide imaging iv. a positive exercise stress test for cardiac ischaemia v. a positive radionuclide exercise, echocardiographic exercise, or pharmacological cardiovascular stress test for cardiac ischaemia vi. coronary revascularization (CABG or PTCA) vii. angiographic evidence of atherosclerotic stenosis > 50% of the diameter of any coronary artery viii. ECG with pathological Q waves in two contiguous leads
   2. heart failure
   3. cerebrovascular disease thought due to atherothrombotic disease
   4. aortic or peripheral vascular disease
   5. or three or more of the following risk factors:

      * age ≥70 years
      * any history of congestive heart failure
      * diabetes and currently on an oral hypoglycaemic agent or insulin therapy
      * current treatment for hypertension
      * preoperative serum creatinine >175 micro mol/L (> 2.0 mg/dl)
      * current or previous high cholesterol ≥6.2 mmol/L (> 240 mg/dl)
      * history of a transient ischemic attack (TIA) (i.e. a transient focal neurological deficit that lasted less than 24 hours and thought to be vascular in origin)
      * emergency/urgent surgery (i.e. surgery which must be undertaken within 24 hours of acute presentation to hospital)
      * high-risk type of surgery (i.e. intrathoracic or intraperitoneal)

Exclusion Criteria

1. having cardiac surgery
2. marked impairment of gas-exchange expected to require Fi02> 0.5 intraoperatively
3. specific circumstances where N2O is contraindicated (eg. volvulus, pulmonary hypertension, raised intracranial pressure) or the anaesthetist plans to use supplemental oxygen (eg. colorectal surgery)
4. N2O unavailable for use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7112 (Actual)
Dates: Start 2007-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Myles, MBBS MPH MD, Principal Investigator — The Alfred
Locations (1):
- Alfred Hosptial, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beattie WS, Wijeysundera DN, Chan MTV, Peyton PJ, Leslie K, Paech MJ, Sessler DI, Wallace S, Myles PS, Galagher W, Farrington C, Ditoro A, Baulch S, Sidiropoulos S, Bulach R, Bryant D, O'Loughlin E, Mitteregger V, Bolsin S, Osborne C, McRae R, Backstrom M, Cotter R, March S, Silbert B, Said S, Halliwell R, Cope J, Fahlbusch D, Crump D, Thompson G, Jefferies A, Reeves M, Buckley N, Tidy T, Schricker T, Lattermann R, Iannuzzi D, Carroll J, Jacka M, Bryden C, Badner N, Tsang MWY, Cheng BCP, Fong ACM, Chu LCY, Koo EGY, Mohd N, Ming LE, Campbell D, McAllister D, Walker S, Olliff S, Kennedy R, Eldawlatly A, Alzahrani T, Chua N, Sneyd R, McMillan H, Parkinson I, Brennan A, Balaji P, Nightingale J, Kunst G, Dickinson M, Subramaniam B, Banner-Godspeed V, Liu J, Kurz A, Hesler B, Fu AY, Egan C, Fiffick AN, Hutcherson MT, Turan A, Naylor A, Obal D, Cooke E; ANZCA Clinical Trials Network for the ENIGMA-II Investigators. Implication of Major Adverse Postoperative Events and Myocardial Injury on Disability and Survival: A Planned Subanalysis of the ENIGMA-II Trial. Anesth Analg. 2018 Nov;127(5):1118-1126. doi: 10.1213/ANE.0000000000003310. PMID 29533264
- [Derived] Corcoran T, Kasza J, Short TG, O'Loughlin E, Chan MT, Leslie K, Forbes A, Paech M, Myles P; ENIGMA-II investigators. Intraoperative dexamethasone does not increase the risk of postoperative wound infection: a propensity score-matched post hoc analysis of the ENIGMA-II trial (EnDEX). Br J Anaesth. 2017 Feb;118(2):190-199. doi: 10.1093/bja/aew446. PMID 28100522
- [Derived] Chan MT, Peyton PJ, Myles PS, Leslie K, Buckley N, Kasza J, Paech MJ, Beattie WS, Sessler DI, Forbes A, Wallace S, Chen Y, Tian Y, Wu WK; and the Australian and New Zealand College of Anaesthetists Clinical Trials Network for the ENIGMA-II investigators. Chronic postsurgical pain in the Evaluation of Nitrous Oxide in the Gas Mixture for Anaesthesia (ENIGMA)-II trial. Br J Anaesth. 2016 Dec;117(6):801-811. doi: 10.1093/bja/aew338. PMID 27956679
- [Derived] Myles PS, Leslie K, Chan MT, Forbes A, Peyton PJ, Paech MJ, Beattie WS, Sessler DI, Devereaux PJ, Silbert B, Schricker T, Wallace S; ANZCA Trials Group for the ENIGMA-II investigators. The safety of addition of nitrous oxide to general anaesthesia in at-risk patients having major non-cardiac surgery (ENIGMA-II): a randomised, single-blind trial. Lancet. 2014 Oct 18;384(9952):1446-54. doi: 10.1016/S0140-6736(14)60893-X. PMID 25142708
- [Derived] Myles PS, Leslie K, Peyton P, Paech M, Forbes A, Chan MT, Sessler D, Devereaux PJ, Silbert BS, Jamrozik K, Beattie S, Badner N, Tomlinson J, Wallace S; ANZCA Trials Group. Nitrous oxide and perioperative cardiac morbidity (ENIGMA-II) Trial: rationale and design. Am Heart J. 2009 Mar;157(3):488-494.e1. doi: 10.1016/j.ahj.2008.11.015. PMID 19249419

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrous Oxide Group: General anaesthesia containing Nitrous oxide and fraction of inspired oxygen of 30%
- No Nitrous Oxide: General anaesthesia not containing Nitrous oxide with fraction of inspired oxygen of 30%
Period: Overall Study
Arm/Group | Nitrous Oxide Group | No Nitrous Oxide
Started | 3543 | 3569
Completed | 3483 | 3509
Not Completed | 60 | 60
Not completed — Lost to Follow-up | 2 | 3
Not completed — Withdrawal by Subject | 15 | 14
Not completed — Protocol Violation | 30 | 37
Not completed — Not eligible | 13 | 6

BASELINE CHARACTERISTICS:
Population: Of 10 102 eligible patients, 7112 patients were enrolled and randomly assigned: 3543 to receive nitrous oxide and 3569 not to receive nitrous oxide; 7011 patients underwent induction of anaesthesia and were included at baseline, and 6992 patients were assessed for the primary endpoint (figure 1).
Groups:
- N2O Group (FiO2 0.3): Nitrous Oxide as an inspired concentration of 70% in 30% Oxygen
- N2O Free Group (FiO2 0.3): Nitrous Oxide free air and inspired Oxygen concentration of 30%
- Total: Total of all reporting groups
Arm/Group | N2O Group (FiO2 0.3) | N2O Free Group (FiO2 0.3) | Total
Number analyzed (Participants) | 3495 | 3516 | 7011
Age, Continuous [Mean (Standard Deviation); unit: years] — AGE>18
  years
    Age | 69.2 (9.8) | 69.5 (9.7) | 69.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1253 | 1299 | 2552
  Male | 2242 | 2217 | 4459
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 706 | 701 | 1407
  Black or African American | 19 | 11 | 30
  White | 2587 | 2630 | 5217
  Other | 13 | 50 | 63
  Indian/Pakistani | 63 | 57 | 120
  Unknown | 107 | 67 | 174

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is a Composite of Death and Cardiovascular Events (Clinical and Silent MI, Cardiac Failure, Cardiac Arrest, Pulmonary Embolism, and Stroke) Measured at 30 Days After Surgery.
Time Frame: 30 days post op
Measure: Number; unit: participants
Groups:
- Nitrous Oxide: 70% N2O (FiO2 0.3): N2O Group (FiO2 0.3)
  Nitrous Oxide: 70% N2O V's No N2O
  Nitrous Oxide: N2O 70% v's No N2O
- N2O Free Group (FiO2 0.3): N2O free group (FiO2 0.3)
  Nitrous Oxide: 70% N2O V's No N2O
  Nitrous Oxide: N2O 70% v's No N2O
Arm/Group | Nitrous Oxide: 70% N2O (FiO2 0.3) | N2O Free Group (FiO2 0.3)
Number analyzed (Participants) | 3483 | 3509
participants | 283 | 296

2. Secondary Outcome: Myocardial Infarction (MI)
Time Frame: 30 days post op
Measure: Number; unit: participants
Arm/Group | Nitrous Oxide: 70% N2O (FiO2 0.3) | N2O Free Group (FiO2 0.3)
Number analyzed (Participants) | 3483 | 3509
participants | 215 | 219

3. Secondary Outcome: Cardiac Arrest
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Nitrous Oxide: 70% N2O (FiO2 0.3) | N2O Free Group (FiO2 0.3)
Number analyzed (Participants) | 3483 | 3509
participants | 15 | 19

4. Secondary Outcome: Pulmonary Embolism
Time Frame: 30 Days Post op
Measure: Number; unit: participants
Groups:
- N2O Group (FiO2 0.3): N2O Group (FiO2 0.3)
- N2O Free Group (FiO2 0.3): N2O free group (FiO2 0.3)
Arm/Group | N2O Group (FiO2 0.3) | N2O Free Group (FiO2 0.3)
Number analyzed (Participants) | 3483 | 3509
participants | 18 | 22

5. Secondary Outcome: Stroke
Time Frame: 30 Days Post op
Measure: Number; unit: participants
Arm/Group | Nitrous Oxide: 70% N2O (FiO2 0.3) | N2O Free Group (FiO2 0.3)
Number analyzed (Participants) | 3483 | 3509
participants | 26 | 19

6. Secondary Outcome: Wound Infection
Time Frame: 30 Days Post op
Measure: Number; unit: participants
Arm/Group | Nitrous Oxide: 70% N2O (FiO2 0.3) | N2O Free Group (FiO2 0.3)
Number analyzed (Participants) | 3483 | 3509
participants | 321 | 311

7. Secondary Outcome: Hospital Stay (Days)
Time Frame: 30 Days Post Op
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Nitrous Oxide: 70% N2O (FiO2 0.3) | N2O Free Group (FiO2 0.3)
Number analyzed (Participants) | 3483 | 3509
Days | 6.1 [3.3 to 10] | 6.1 [3.3 to 10]

ADVERSE EVENTS:
Time Frame: 30 Days
Description: Adverse events do not include the primary endpoint variables
Groups:
- Nitrous Oxide: 70% N2O: N2O Group (FiO2 0.3)
  Nitrous Oxide: 70% N2O V's No N2O
  General anaesthesia containing Nitrous oxide and fraction of inspired oxygen of 30%
- Nitrous Oxide Free: Nitrous Oxide free group (FiO2 0.3)
  Nitrous Oxide: N2O 70% v's No N2O
  General anaesthesia not containing Nitrous oxide and fraction of inspired oxygen of 30%
Arm/Group | Nitrous Oxide: 70% N2O | Nitrous Oxide Free
All-Cause Mortality (participants affected / at risk) | 42/3483 | 57/3509
Serious Adverse Events (participants affected / at risk) | 283/3483 | 296/3509
Other Adverse Events (participants affected / at risk) | 662/3483 | 546/3509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrous Oxide: 70% N2O (N=3483) | Nitrous Oxide Free (N=3509)
Myocardial Infarction (Cardiac disorders) | 215 (215) | 219 (219)
Stroke (Blood and lymphatic system disorders) | 26 (26) | 19 (19)
Cariac Arrest (Cardiac disorders) | 15 (15) | 19 (19)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 22 (22)
Death (General disorders) | 42 (42) | 57 (57)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitrous Oxide: 70% N2O (N=3483) | Nitrous Oxide Free (N=3509)
Neurological (Nervous system disorders) | 53 (53) | 48 (48)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 103 (103) | 93 (93)
Gastrointestinal (Gastrointestinal disorders) | 106 (106) | 85 (85)
Cardiovascular (Cardiac disorders) | 90 (90) | 25 (25)
Urology (Renal and urinary disorders) | 72 (72) | 73 (73)
Vascular (Vascular disorders) | 50 (50) | 38 (38)
Bleeding complications (Blood and lymphatic system disorders) | 54 (54) | 56 (56)
Other (Investigations) | 134 (134) | 128 (128) — All other events less than 2% overall

LIMITATIONS AND CAVEATS:
All 'other' adverse events the events were classed according to system MedDRA reporting and not by individual event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes